CLINICAL TRIAL: NCT02899338
Title: Randomized, Single-dose, Parallel-arm, Open-label Phase I Trial to Compare the Pharmacokinetics, Safety and Tolerability of BI 695501 Administered Subcutaneously Via Prefilled Syringe or Autoinjector
Brief Title: Pharmacokinetics and Safety of BI 695501
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1297.13; 2016-003158-34 (EudraCT Number)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Healthy

ARMS (2):
- BI695501 Autoinjector (Experimental)
  Interventions: Drug: BI695501Autoinjector
- BI695501 Prefilled syringe (Active Comparator)
  Interventions: Drug: BI695501 Prefilled syringe

INTERVENTIONS:
Drug: BI695501 Prefilled syringe
  Arms: BI695501 Prefilled syringe
Drug: BI695501Autoinjector
  Arms: BI695501 Autoinjector

SUMMARY:
To characterize and compare the pharmacokinetics and to assess the safety of BI 695501 after single injection using either auto injector or prefilled syringe.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 65 years (inclusive)
* BMI of >17.5 to <35.0 kg/m2
* Healthy male or female subjects, according to the investigator´s assessment, based on a complete medical history including a physical examination, vital signs (blood pressure [BP], pulse rate [PR]), 12-lead ECG, and clinical laboratory tests.
* Subjects who meet any of the following criteria:

  * Surgically sterilized (confirmed 6 month prior to enrollment)
  * Have surgically sterilized sexual partner (confirmed 6 month prior to enrollment)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)
* Subjects agree to use an adequate contraception, starting from the begin of the trial and until 6 months after the dose of the trial drug: e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the trial

Exclusion criteria:

* Previous exposure to adalimumab or proposed adalimumab biosimilar drugs.
* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) that deviates from normal and judged as clinically relevant by the investigator.
* Any evidence of a concomitant disease judged as clinically relevant by the investigator including gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal disorders or diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension, fainting spells, or blackouts.
* Chronic or relevant acute infections.
* Positive result for HIV, hepatitis B virus (HBV), and hepatitis C (Hep C) at screening.
* History of relevant allergy or hypersensitivity including allergy to the trial medication, its excipients or device materials (e.g. natural rubber or latex).
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial.
* Intake of an investigational drug in another trial within 2 months or 5 half-lives (whichever longer) prior to planned administration of the trial medication in this trial or intake of an investigational drug during the course of this trial.
* Alcohol abuse (consumption of more than 28 units/week).
* Unwillingness/inability to refrain from intake of alcoholic beverages from 48 hours prior to the trial medication administration and until Day 14 post trial medication administration; and/or to limit alcohol intake to a maximum of 3 units per day until e.o.t.
* Drug abuse or positive drug screening.
* Blood donation of more than 500 mL within 30 days prior to administration of trial medication or intended donation during the trial.
* Intention to perform excessive physical activities within 4days prior to administration of trial medication or contact sport during the entire trial and unwilling to avoid vigorous exercise for 14 days post dosing.
* Inability to comply with dietary regimen of trial site.
* Any out-of-range laboratory values considered clinically significant by the investigator; (subjects with creatine kinase (CK) values 2 times the upper limit of normal (ULN) at Day -1 are to be excluded from participation).
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because he is considered not able to understand and comply with trial requirements, or has a condition that would not allow safe participation in the trial.
* Subjects with any immunological disorders or auto-immune disorders, (e.g., Rheumatoid arthritis (RA), lupus erythematosus, scleroderma, etc.).
* Subject has received a live vaccine within 12 weeks prior to enrolling in the trial.
* History of tuberculosis (TB) or positive finding in Interferon-gamma release assay (IGRA).
* Evidence of skin irritation or infection at the planned injection place.
* Currently enrolled in another investigational device or drug study
* Any condition that, in the investigator´s opinion, makes them an unreliable study subject or unlikely to complete the trial
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- SGS Life Sciences Services, Antwerp, Belgium
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized in 1:1 ratio to receive BI 695501 (autoinjector) or BI 695501 (prefilled syringe).
Groups:
- BI695501 Prefilled Syringe: Patients were administered a single subcutaneous dose of 40 milligram (mg)/0.8 milliliter (mL) BI 695501 (solution for injection) using a prefilled syringe (PFS).
- BI695501 Autoinjector: Patients were administered a single subcutaneous dose of 40 milligram (mg)/0.8 milliliter (mL) BI 695501 (solution for injection) using an autoinjector (AI).
Period: Overall Study
Arm/Group | BI695501 Prefilled Syringe | BI695501 Autoinjector
Started | 81 | 81
Completed | 78 | 79
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | BI695501 Prefilled Syringe | BI695501 Autoinjector | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] — Mean (SD) of age at enrollment is presented.
  Years | 44.5 (14.74) | 41.5 (14.44) | 43.0 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects are presented as male/female in each treatment group.
  Participants
    Female | 44 | 43 | 87
    Male | 37 | 38 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects having different ethnicities are presented.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 81 | 81 | 162
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects belonging to different races are presented.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 1 | 4
    White | 78 | 77 | 155
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1
Body weight at baseline [Mean (Standard Deviation); unit: Kilogram (kg)] — Body weight at baseline is presented.
  Kilogram (kg) | 74.84 (15.421) | 75.25 (14.909) | 75.04 (15.122)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 695501 in Plasma Over the Time Interval From 0 to 1368 Hours (AUC0-1368) After Administration Via PFS and AI.
Description: The AUC0-1368 of 40 mg BI 695501 administered via PFS and AI was measured. Plasma concentrations were measured using a validated enzyme-linked immunosorbent assay (ELISA). Only concentration values within the validated concentration range of 0.025 to 2.0 micrograms per millilitre (µg/mL) and actual sampling times were used.
Time Frame: From 0 to 1368 hours post-dose. Samples were collected pre-dose and 1, 4, 8, 12, 24, 48, 60, 72, 84, 96, 108, 120, 132, 144, 168, 216, 336, 504, 672, 840, 1032, and 1368 hours post-dose.
Population: PKS: The pharmacokinetic set (PKS) consisted of all randomized subjects who received the single dose of trial medication (BI 695501 administered via PFS or AI), had at least 1 evaluable primary PK parameter, and were without important protocol deviations or violations thought to significantly affect the PK of BI 695501.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram hour per milliliter (μg*h/mL)
Arm/Group | BI695501 Prefilled Syringe | BI695501 Autoinjector
Number analyzed (Participants) | 76 | 79
microgram hour per milliliter (μg*h/mL) | 2100 (43.9) | 2150 (45.2)
Statistical Analysis 1: Comparison: BI695501 Prefilled Syringe vs BI695501 Autoinjector; Comparison AI versus PFS; Test type: Equivalence — The relative bioavailability of BI 695501 using AI (A) compared with BI 695501 using PFS (B) was estimated, in an exploratory manner, by the ratios of the geometric means (A/B) using the analysis of variance (ANOVA); ANOVA; The results are based on ANOVA model on the logarithmic scale with fixed effects for treatment and baseline body weight; Adjusted geometric mean ratio = 101.71, 90% CI 2-sided [91.31 to 113.29], Standard Error of Mean 42.28 — Standard error of the mean is actually the Inter-individual geometric coefficient of variation (gCV)

2. Primary Outcome: The Maximum Measured Concentration of BI 695501 in Plasma (Cmax) After Administration Via PFS and AI
Description: The Cmax of 40 mg BI 695501 administered via PFS and AI. Plasma concentrations were measured using a validated ELISA. Only concentration values within the validated concentration range of 0.025 to 2.0 µg/mL and actual sampling times were used.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | BI695501 Prefilled Syringe | BI695501 Autoinjector
Number analyzed (Participants) | 79 | 81
µg/mL | 3.86 (27.8) | 3.86 (23.6)
Statistical Analysis 1: Comparison: BI695501 Prefilled Syringe vs BI695501 Autoinjector; Comparison AI versus PFS; Test type: Equivalence — The relative bioavailability of BI 695501 using AI (A) compared with BI 695501 using PFS (B) was estimated, in an exploratory manner, by the ratios of the geometric means (A/B) using ANOVA; ANOVA; The results are based on ANOVA model on the logarithmic scale with fixed effects for treatment and baseline body weight; Adjusted geometric mean ratio = 100.11, 90% CI 2-sided [94.17 to 106.43], Standard Error of Mean 23.72 — Standard error of the mean is actually the Inter-individual gCV

3. Primary Outcome: Area Under the Concentration-time Curve of BI 695501 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞) After Administration Via PFS and AI.
Description: The AUC0-∞ of 40 mg BI 695501 administered via PFS and AI. Plasma concentrations were measured using a validated ELISA. Only concentration values within the validated concentration range of 0.025 to 2.0 µg/mL and actual sampling times were used.
Time Frame: Samples were collected pre-dose and 1, 4, 8, 12, 24, 48, 60, 72, 84, 96, 108, 120, 132, 144, 168, 216, 336, 504, 672, 840, 1032, and 1368 hours post-dose.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | BI695501 Prefilled Syringe | BI695501 Autoinjector
Number analyzed (Participants) | 76 | 79
μg*h/mL | 2250 (50.3) | 2330 (50.4)
Statistical Analysis 1: Comparison: BI695501 Prefilled Syringe vs BI695501 Autoinjector; Comparison AI versus PFS; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; The results are based on ANOVA model on the logarithmic scale with fixed effects for treatment and baseline body weight; Adjusted geometric mean ratio = 103.19, 90% CI 2-sided [91.38 to 116.53], Standard Error of Mean 48.21 — Standard error of the mean is actually the Inter-individual gCV

4. Secondary Outcome: The Percentage of Subjects With Drug-related Treatment-emergent Adverse Events (TEAEs) From Day 1 to Day 70.
Description: A treatment-related TEAE was defined as any TEAE assessed by the Investigator as related to the trial medication. A TEAE was defined as an adverse event (AE) that started or worsened in severity on or after the single dose of trial medication up to 10 weeks (70 days) post-dose.
Time Frame: From Day 1 to Day 70
Population: All treated subjects (i.e. all subjects who received 1 dose of trial medication) were included in the safety analysis set (SAF).
Measure: Number; unit: Percentage of participants
Arm/Group | BI695501 Prefilled Syringe | BI695501 Autoinjector
Number analyzed (Participants) | 81 | 81
Percentage of participants | 37.0 | 38.3

ADVERSE EVENTS:
Time Frame: From single dose administration till 10 weeks; up to 70 days
Description: All events with an onset after the single dose of trial medication up to a period of 10 weeks (70 days) were assigned to the treatment phase for evaluation and were considered to be TEAEs. The SAF population was used which consisted of all subjects that received a single dose of trial medication.
Arm/Group | BI695501 Autoinjector | BI695501 Prefilled Syringe
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81
Serious Adverse Events (participants affected / at risk) | 2/81 | 1/81
Other Adverse Events (participants affected / at risk) | 47/81 | 41/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI695501 Autoinjector (N=81) | BI695501 Prefilled Syringe (N=81)
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI695501 Autoinjector (N=81) | BI695501 Prefilled Syringe (N=81)
Abdominal discomfort (Gastrointestinal disorders) | 8 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 8 | 4
Influenza like illness (General disorders) | 5 | 5
Injection site erythema (General disorders) | 14 | 7
Injection site haematoma (General disorders) | 6 | 0
Injection site induration (General disorders) | 4 | 5
Injection site pain (General disorders) | 5 | 4
Injection site swelling (General disorders) | 6 | 5
Nasopharyngitis (Infections and infestations) | 11 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Headache (Nervous system disorders) | 16 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT02899338/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT02899338/SAP_001.pdf